CLINICAL TRIAL: NCT03862742
Title: Role of Wrist Based Blood Pressure Monitoring in Clinical Practice
Status: Withdrawn | Type: Observational
Why Stopped: No participants enrolled.
Sponsor: Scripps Translational Science Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-18-7223
Record Dates: First submitted 2019-02-21; First posted 2019-03-05 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure; Transitions of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients admitted to the hospital: We will recruit patient volunteers from the Scripps Green Hospital and Scripps Memorial Hospital inpatient teaching services.

SUMMARY:
This is a pilot clinical study to test the overarching hypothesis that frequent and longitudinal blood pressure monitoring with FDA approved consumer wrist based device during the patient transition from inpatient to home to the first clinic visit will elicit valuable BP data that can assist in physician treatment of hypertension

DETAILED DESCRIPTION:
Wrist based health devices, often with mobile connectivity, that continuously or near continuously track heart rate, blood pressure, temperature, activity and sleep are growing in everyday popularity and beginning to enter the sphere of clinical relevance. However, their accuracy and utility for clinical use is largely unstudied. As these consumer devices, some of which are FDA approved, become more commonplace, it is paramount to understand their function, know their limitations, and be able to interpret results appropriately before incorporating them into our clinical practice. The AHA/ACC 2017 guideline makes a 1A recommendation for clinical use of out of office BP measurements(1). This recommendation is based on evidence that out of office BP and frequent and longitudinal BP measurements are important in predicting cardiovascular risk and monitoring treatment efficacy(2-5). This trend towards consumer driven digital health monitoring and the new AHA/ACC guideline are essentially advancing a consumer based precision medicine strategy for diagnosis and monitoring of hypertension. As this becomes commonplace in our patient population, we need rigorous clinical study of wrist base BP monitoring to better understand its role patient care.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Own an iOS or Android device

Exclusion Criteria:

* Inability to give informed consent
* <18 years of age
* Inability to understand written English language
* Hypertensive urgency or emergency as an admission diagnosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals 18 years of age or older with and without the known diagnosis of hypertension (regardless of level of control or therapeutic regimen), able to operate HeartVue device, able to read, write, and speak English, level of "digital savviness" and owning an iOS or Android device will be recruited for participation in this pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Pts will monitor BP during the transition from inpatient to home to the first clinic visit. BP measurements will be performed several times during the day and several times at night. The estimated time frame when data will be collected is 24 to 48 hours
  blood pressure measured by the wrist watch like blood pressure device

SECONDARY OUTCOMES:
Survey of healthcare providers | A survey to measure how easy it is to use the device will be obtained at the completion of data collection. The estimated timeframe when the survey will be completed is 24 to 48 hours.
  Survey to measure ease of use to the device in measuring blood pressure
Survey of patients | A survey to measure how easy it is to use the device will be obtained at the completion of data collection. The estimated timeframe when the survey will be completed is 24 to 48 hours.
  Survey to measure ease of use to the device in measuring blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Laura Nicholson, MD PHD, Principal Investigator — Scripps Health
Locations (1):
- Scripps Green Hospital, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. J Am Soc Hypertens. 2018 Aug;12(8):579.e1-579.e73. doi: 10.1016/j.jash.2018.06.010. No abstract available. PMID 30219548
- [Background] Drawz P. Clinical Implications of Different Blood Pressure Measurement Techniques. Curr Hypertens Rep. 2017 Jul;19(7):54. doi: 10.1007/s11906-017-0751-0. PMID 28551831
- [Background] O'Brien E, Parati G, Stergiou G, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring. European Society of Hypertension position paper on ambulatory blood pressure monitoring. J Hypertens. 2013 Sep;31(9):1731-68. doi: 10.1097/HJH.0b013e328363e964. PMID 24029863
- [Background] Hermida RC, Ayala DE, Fernandez JR, Mojon A, Smolensky MH. Hypertension: New perspective on its definition and clinical management by bedtime therapy substantially reduces cardiovascular disease risk. Eur J Clin Invest. 2018 May;48(5):e12909. doi: 10.1111/eci.12909. Epub 2018 Feb 25. PMID 29423914
- [Background] Staessen JA, Thijs L, Fagard R, O'Brien ET, Clement D, de Leeuw PW, Mancia G, Nachev C, Palatini P, Parati G, Tuomilehto J, Webster J. Predicting cardiovascular risk using conventional vs ambulatory blood pressure in older patients with systolic hypertension. Systolic Hypertension in Europe Trial Investigators. JAMA. 1999 Aug 11;282(6):539-46. doi: 10.1001/jama.282.6.539. PMID 10450715

DOCUMENTS (2):
  • Study Protocol (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03862742/Prot_002.pdf
  • Statistical Analysis Plan (2018-10-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03862742/SAP_003.pdf